CLINICAL TRIAL: NCT03733496
Title: An Observational, Long-Term Extension Study for Participants in Prior VY-AADC01 Clinical Studies
Brief Title: Observational, Long-term Extension Study for Participants of Prior VY-AADC01 Studies
Status: Completed | Type: Observational
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Voyager Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-1104
Record Dates: First submitted 2018-10-19; First posted 2018-11-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease (PD); Gene Therapy; Motor Fluctuations; Neurosurgery; NBIb-1817; Aromatic L-Amino Acid Decarboxylase; Levodopa; Dopamine; AADC; DDC; AAV2-hAADC; AAV; VY-AADC
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from VY-AADC01 clinical studies:: Participants who have completed participation in VY-AADC01 clinical studies (PD-1101 or PD-1102) will be invited to participate in this extension study

SUMMARY:
An extension study for participants who have completed a prior VY-AADC01 clinical study

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed participation in the PD-1101 or PD-1102 clinical study of VY-AADC01 gene therapy

Key Exclusion Criteria:

None

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants from prior VY-AADC01 clinical studies will be eligible for the extension study
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 8 years from VY-AADC01 administration
  Long-term safety of VY-AADC01 as measured by Adverse Events and Serious Adverse Events

SECONDARY OUTCOMES:
Change in AADC enzyme activity | Up to 8 years from VY-AADC01 administration
  Continued expression of AADC as measured by [18F]-fluorodopa (F-Dopa) positron emission tomography (PET)
Changes in PD medications | Up to 8 years from VY-AADC01 administration
  Change from baseline in PD medications, measured as levodopa equivalent dose
Changes in motor function as assessed by Unified Parkinson's Disease Rating Scale (UPDRS) | Up to 8 years from VY-AADC01 administration
  Changes from baseline in motor function as assessed by UPDRS, in both "Off" and "On" medication states
Changes in "Off" and "On" time as recorded by the participant in Parkinson's Disease (PD) diary | Up to 8 years from VY-AADC01 administration
  Changes from baseline based on the PD Diary: "OFF" time; "ON" time without troublesome dyskinesia; "ON" time without dyskinesia; "ON" time with troublesome dyskinesia; and "ON" time with non-troublesome dyskinesia

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christine CW, Bankiewicz KS, Van Laar AD, Richardson RM, Ravina B, Kells AP, Boot B, Martin AJ, Nutt J, Thompson ME, Larson PS. Magnetic resonance imaging-guided phase 1 trial of putaminal AADC gene therapy for Parkinson's disease. Ann Neurol. 2019 May;85(5):704-714. doi: 10.1002/ana.25450. Epub 2019 Mar 26. PMID 30802998
- [Background] Richardson RM, Bankiewicz KS, Christine CW, Van Laar AD, Gross RE, Lonser R, Factor SA, Kostyk SK, Kells AP, Ravina B, Larson PS. Data-driven evolution of neurosurgical gene therapy delivery in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2020 Nov;91(11):1210-1218. doi: 10.1136/jnnp-2020-322904. Epub 2020 Jul 30. PMID 32732384
- [Background] Nutt JG, Curtze C, Hiller A, Anderson S, Larson PS, Van Laar AD, Richardson RM, Thompson ME, Sedkov A, Leinonen M, Ravina B, Bankiewicz KS, Christine CW. Aromatic L-Amino Acid Decarboxylase Gene Therapy Enhances Levodopa Response in Parkinson's Disease. Mov Disord. 2020 May;35(5):851-858. doi: 10.1002/mds.27993. Epub 2020 Mar 9. PMID 32149427